CLINICAL TRIAL: NCT05434741
Title: Feasibility and Acceptability of a Cognitive Behavioral Therapy (CBT)-Based Group Intervention to Reduce Inflammation in Older People With HIV
Brief Title: Cognitive Behavior Therapy (CBT)-Based Group Intervention to Reduce Inflammation in Older People With HIV
Acronym: CHAMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Abigail Batchelder, Ph.D., M.P.H., Principal Investigator, Assistant Professor, Staff Psychologist, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2022P001224; 2022A000527 (Other Grant/Funding Number: The Mongan Institute)
Record Dates: First submitted 2022-06-17; First posted 2022-06-28 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2024-12

CONDITIONS: Aging; HIV

STUDY DESIGN:
Intervention Model Description: This study is a pilot randomized controlled trial, which will include 50 older people with HIV. Each block (n = 4) will be 1:1 randomized to either the group intervention or information-only control.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBT Group (Experimental): This 12-week intervention program leverages evidence-based traditional and contemporary CBT strategies, with the goal of improving the psychological and physical functioning of older people with HIV by providing education and support to learn strategies to: a.) better manage stressors associated with HIV and aging (e.g., treatment access and engagement, and multi-morbidity), and b.) increase health-promoting behaviors (e.g., physical activity).
  Interventions: Behavioral: Weekly Group Skills
- Information-only Group (Experimental): Participants in the control group will receive a one-time trifold brochure titled "HIV: 50 Years or Older."
  Interventions: Other: One-time Trifold Brochure titled "HIV: 50 Years or Older"

INTERVENTIONS:
Behavioral: Weekly Group Skills — The topics covered in group CBT sessions are: 1.) Domains of Healthy Aging; 2.) Stress and anxiety; 3.) Adherence and Engagement in Primary/Preventative Care; 4.) Depression and Distress; 5.) Physical Activity; 6.) Stigma/Self-Compassion; 7.) Substance Use; 8.) Acceptance of Uncertainty and Uncomfortable Emotions; 9.) Diet; 10.) Behavioral Activation; 11.) Frailty and Memory/Cognition; and 12.) Wrap-Up and Maintaining Gains.
  Arms: CBT Group
Other: One-time Trifold Brochure titled "HIV: 50 Years or Older" — Participants in the education only group will receive a one-time trifold brochure titled "HIV: 50 Years or Older. This brochure contains information on the prevalence of HIV among people aged 50 and older, defines medication adherence and drug resistance, encourages physical activity and proper nutrition, and addresses the health risk behavior of tobacco-smoking for people living with HIV. Participants receive one brochure in the information-only group.
  Arms: Information-only Group

SUMMARY:
In this study, the investigators will assess the feasibility and acceptability of an evidence-based CBT group intervention, developed for older people with HIV, and research methods in a pilot randomized controlled trial including 50 older people with HIV as participants. The evidence-based CBT intervention has been developed and utilized in three clinical groups to date initiated and led by Dr. Batchelder (PI) in the Behavioral Medicine program at MGH. The 12-week intervention program proposed leverages evidence-based traditional and contemporary CBT strategies, with the goal of improving the psychological and physical functioning of older people with HIV by providing education and support to learn strategies to: a.) better manage stressors associated with HIV and aging (e.g., multi-morbidity), and b.) increase health-promoting behaviors (e.g., physical activity).

DETAILED DESCRIPTION:
This study is a pilot randomized controlled trial, which will include 50 older people with HIV as participants. Blocks (n = 4) will be 1:1 randomized to either the group intervention or information-only control. The established 12-week group intervention consists of evidence-based traditional and contemporary CBT strategies. Each week will focus on a distinct theme, including: 1.) Domains of Healthy Aging; 2.) Stress and anxiety; 3.) Adherence and Engagement in Primary/Preventative Care; 4.) Depression and Distress; 5.) Physical Activity; 6.) Stigma/Self-Compassion; 7.) Substance Use; 8.) Acceptance of Uncertainty and Uncomfortable Emotions; 9.) Diet; 10.) Behavioral Activation; 11.) Frailty and Memory/Cognition; and 12.) Wrap-Up and Maintaining Gains.

All participants, including those in the intervention group and in the education-only group, will attend virtual baseline and follow-up appointments, complete computerized self-report measures (REDCap) at baseline and follow-up, a structured diagnostic interview at baseline, and a blood draw appointment at baseline and follow-up. Participants in the education-only group will receive a one-time brochure with information on living with HIV, healthy aging, and healthy behaviors when they attend the baseline blood draw appointment.

Aim 1: Assess the feasibility and acceptability of an evidence-based CBT group intervention, developed for older people with HIV, and research methods in a pilot randomized controlled trial (RCT).

Aim 2: Explore changes in a.) inflammation biomarkers (i.e., interleukin-6 [IL-6] and C-reactive protein [CRP]), b.) psychological distress (i.e., general distress, HIV-specific stress, and depressive and anxiety symptoms), and c.) health risk behaviors (i.e., tobacco-smoking, alcohol use, sedentary behaviors, and poor diet quality) in the intervention group versus an education-only group.

ELIGIBILITY:
Inclusion Criteria:

* HIV+ with an undetectable test result within the last 12 months; willing to provide printed or online version of test result for confirmation
* 50 years of age or older
* On effective ART; willing to provide ART-related health records or prescriptions for confirmation
* Fluent in English (speaking and reading)
* Willing and able to provide informed consent
* Psychiatrically stable based on clinical interview

Exclusion Criteria:

-HIV-

* Unable to provide undetectable HIV test result within the last 12 months
* Not on effective ART
* <50 years old
* Unable to read and write in English
* Unable to provide informed consent

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-06-20 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Acceptability of the CBT group intervention | 12-week follow-up
  Acceptability will be assessed with a satisfaction evaluation survey previously used with similar samples, modeled after the Client Satisfaction Questionnaire (CSQ-8).
Feasibility of the CBT group intervention | 12-week follow-up
  Feasibility data will consist of attendance patterns. Feasibility of assessment will be the completion of at least 75% of scheduled group sessions.

SECONDARY OUTCOMES:
Changes in psychological distress | Baseline and at 12-week follow-up appointments.
  Investigators will administer the General Distress Screener - K10. Scores range from 10-50 and higher scores indicate greater likelihood of mental illness.
Feasibility of the CBT intervention | 12-week follow-up
  Feasibility data will consist of effort required to recruit the sample (e.g., number of staff members).
Feasibility of the CBT intervention | 12-week follow-up
  Feasibility data will consist of numbers of screenings conducted.
Feasibility of the CBT group intervention | 12-week follow-up
  Feasibility data will consist of the proportion of the sample eligible to participate to participants who agree to enroll. Feasibility of recruitment will be an enrollment rate equal to or greater than 70% of those who are eligible.
Acceptability of the CBT group intervention | Weekly
  Investigators will administer weekly surveys to assess acceptability among participants in the group skills intervention. This survey consists of 4 items assessing content perception.

CONTACTS AND LOCATIONS:
Locations (1):
- One Bowdoin Square, Floor 7, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No